CLINICAL TRIAL: NCT01954160
Title: Promotion of Renal Sodium Excretion by Renal Sympathetic Denervation in Congestive Heart Failure
Brief Title: Study of Renal Denervation in Patients With Heart Failure
Acronym: PRESERVE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMB decision based upon noted lack of efficacy in manufacturers pivotal trials.
Sponsor: Adrian Hernandez (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Adrian Hernandez, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00047050; 5U10HL084904 (NIH)
Record Dates: First submitted 2013-09-24; First posted 2013-10-01 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2015-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Symplicity Renal Denervation (Other): Subjects undergo Symplicity Renal Denervation within 2 weeks of baseline visit will follow usual care after week 13 visit
  Interventions: Device: Symplicity Renal Denervation
- Late Symplicity Renal Denervation (Other): Subjects following usual care until week 13 visit will then undergo Symplicity Renal Denervation within 2 weeks of Week 13 visit
  Interventions: Device: Symplicity Renal Denervation

INTERVENTIONS:
Device: Symplicity Renal Denervation — Renal denervation

SUMMARY:
Congestive heart failure is a common disorder in which the heart cannot pump enough blood to meet the needs of the rest of the body. Poor sodium handling by the kidneys is a damaging effect of heart failure, and it leads to symptoms of congestion such as shortness of breath or ankle swelling. Recent studies suggest that reducing the nerve activity to a kidney could reduce sodium retention and blood pressure. An improvement in the way the kidneys handle sodium may reduce disease progression and decrease symptoms for heart failure patients.

DETAILED DESCRIPTION:
Over the past decades, clinical trials in HF have been unable to alter the natural history of cardio-renal compromise. Fluid retention accounts for the majority of admissions for acute decompensated heart failure, and salt and water removal using intravenous (IV) diuretics has been the mainstay of therapy applied to this population.1 Over 20% of hospitalized patients in the Acute Decompensated Heart Failure National Registry (ADHERE) had serum creatinine values greater than 2.0 mg/dL2 with the majority of congested patients presenting with significantly elevated systolic blood pressures rather than low-output states.1 Administration of IV loop diuretics further produces intravascular volume depletion and reduction in glomerular filtration rates3 as well as an increase in neurohormonal activation.4 This is true regardless of whether LVEF is impaired or preserved.5 However, despite relieving symptoms, acute drug administrations (such as adenosine receptor antagonists or natriuretic peptide analogues) for short durations have not changed the long-term cardio-renal outcomes in large clinical trials.

Recent recognition of different phenotypes of cardio-renal syndrome has provided better characterization of patient populations to evaluate specific treatment approaches or interventions.6 There is now greater appreciation that patients with congestive HF depend not only on an adequate glomerular function for renal glomerular filtration, but also on adequate tubular function for effective sodium handling that may or may not be dependent on glomerular filtration.7 Despite optimizing intracardiac filling pressures, many patients with August 28, 2013 Page 10 of 58 cardio-renal compromise remain symptomatic, complaining of breathlessness and fatigue often associated with concomitant increase in neurohormonal up-regulation (e.g. natriuretic peptides) and poor outcomes.8 Since the majority of patients present with hypertension, it points to the possibility that congestive HF is precipitated by heightened sympathetic drive.

Animal models have demonstrated that both blood pressure control and renal tubular function/glomerular filtration (as a function of renal blood flow) can be directly influenced by renal sympathetic nerve activity,9-12 which has evolved to provide cardiovascular support in the setting of hypovolemia or profound cardiovascular collapse. Specifically, HF animal models with denervated kidneys have demonstrated improvement in renal blood flow and natriuresis (with restoration of Na+-K+ ATPase at the loop of Henle, as well as epithelial sodium pumps at the distal tubules). However, our understanding of how persistently activated renal sympathetic outflow can lead to exaggerated neurohormonal up-regulation and chemoreceptor regulation in humans is still evolving. As heightened cardio-renal compromise leads to disease progression and congestive HF, it is conceivable that an approach to selectively modulate renal sympathetic outflow may improve cardio-renal compromise as well as the target mechanism leading to symptomatic improvement in at-risk patients.

By establishing the mechanistic role of renal sympathetic outflow in patients with impaired sodium handling as a contributor to congestion in HF, we may better understand why patients with HF develop symptoms, retain salt and water, and activate neurohormonal systems. This trial will be hypothesis generating and will serve to inform a larger clinical trial in patients with congestion related to HF.

The Data Safety and Monitoring Board (DSMB), an independent committee assigned by the sponsor to oversee the conduct and safety of this study, met on May 12, 2014 to review information that had become available from another study of the renal artery denervation procedure using the same investigational catheter as the PRESERVE study. Even though there were no concerns for the safety of subjects that had the renal artery denervation, the DSMB decided to stop the PRESERVE study.

Based upon agreement with the FDA, the protocol was amended to reduce subject participation from 52 weeks to 13 weeks and to only collect limited safety information.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 21-80 years old.
* History of chronic HF (>6 months) with current NYHA II-III symptoms.
* Left Ventricular Ejection Fraction ≤40% on a clinically indicated echocardiogram obtained within 6 months prior to informed consent.
* Requires daily loop diuretic (≥40mg furosemide per day, or equivalent) to maintain euvolemia (absence of congestive signs including jugular venous distension with Jugular Venous Pressure > 7cm H20, ≥ moderate (2+) peripheral edema, S3).
* Optimized medical therapy for HF. Patients will be receiving guideline-recommended therapy (per the 2013 ACCF/AHA HF Guidelines) including angiotensin-converting enzyme (ACE) inhibitors and/or angiotensin receptor blocker, beta-blockers, and aldosterone antagonists without changes in heart failure medication regimen (including diuretics) for previous 14 days.
* Systolic blood pressure (BP) ≥110 mmHg at time of informed consent.
* Able to maintain stable medications for 52 weeks.
* Suitable renal artery anatomy for Renal Sympathetic Denervation (RSD) procedure. All of the following criteria must be met, based on the screening renal Doppler ultrasound:
* ≥ 20mm treatable length in each renal artery,
* Diameter in treatable segments must be ≥4mm,
* Lone main renal vessel feeding each kidney.

Exclusion Criteria:

* Unable to comply with protocol or procedures.
* Evidence of orthostatic hypotension or known dysautonomia. Orthostatic hypotension is defined by ≥1 of the following feature(s) within 2-5 minutes of quiet standing:
* ≥ 20 mmHg fall in systolic pressure
* ≥ 10 mmHg fall in diastolic pressure
* Symptoms of cerebral hypoperfusion (e.g. dizziness or lightheadedness, visual blurring or darkening of the visual fields, syncope).
* Evidence of or history of renal artery stenosis, nephrectomy, or renal transplant.
* Significant renal impairment as defined by estimated glomerular filtration rate (eGFR) < 45 ml/min/1.73m2 determined by Modification of Diet in Renal Disease (MDRD) equation.
* Significant proteinuria (>2g protein/daily protein excretion).
* Body mass index (BMI) >35 kg/m2.
* Acute coronary syndrome within last 4 weeks as defined by ECG changes and biomarkers of myocardial necrosis (e.g. troponin) in an appropriate clinical setting (chest discomfort or angina equivalent).
* Coronary revascularization procedures (percutaneous coronary intervention or cardiac artery bypass graft) and or valve surgery within 30 days of screening or expected procedures within the next 6 months.
* Cardiac resynchronization therapy, with or without implantable cardiac defibrillator within 90 days of screening or expected procedures within the next 6 months.
* Hypertrophic or restrictive cardiomyopathy, constrictive pericarditis, active myocarditis, active endocarditis, or complex congenital heart disease.
* Severe advanced HF, with ANY of the following features:
* Current or anticipated use of ventricular assist device within the next 6 months.
* Current or anticipated IV vasoactive drug therapy for HF management within the next 6 months.
* Listed cardiac transplant candidate, with transplantation likely within the next 6 months.
* Known allergic reactions to iodinated radiological contrast media or iodinated antiseptics.
* Greater than moderate mitral or aortic stenosis, and/or severe tricuspid regurgitation.
* Terminal illness (other than HF) with expected survival of less than 1 year.
* Female who is pregnant, nursing, or of childbearing potential not practicing effective birth control.
* Enrollment or planned enrollment in another clinical trial within the next 12 months.
* History of urinary outflow tract obstruction, bladder retention and/ or moderate to severe prostate hypertrophy.
* History of adrenal insufficiency
* History of untreated hypothyroidism
* Patients with non-cardiac dyspnea or fatigue due to frailty, motivational factors, pulmonary disease or orthopedic problems that precludes them from performing 6MWT (Six-Minute WalkTest).

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hernandez, MD, Principal Investigator — Duke University; Eugene Braunwald, MD, Study Chair — Harvard University
Locations (12):
- United States (12):
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Metro Health System, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - The University of Vermont - Fletcher Allen Health Care, Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants were enrolled. 4 subjects received treatment, 1 subject did not receive treatment due to ineligibility secondary to renal doppler findings.
Groups:
- Early Renal Denervation: Subjects undergo renal denervation within 2 weeks of baseline visit
  Symplicity Renal Denervation System
- Late Renal Denervation: Subjects undergo renal denervation within 2 weeks of Week 13 visit
  Symplicity Renal Denervation System
Period: Overall Study
Arm/Group | Early Renal Denervation | Late Renal Denervation
Started | 5 | 0 (Not started)
Completed | 0 (Only 4 subjects completed the first early denervation. No subjects completed the late denervation.) | 0
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Population: All patients were required to have suitable anatomy per renal ultrasound. One randomized subject did not have suitable anatomy to proceed to renal denervaton.
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Renal Denervation | Late Renal Denervation | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 4 |  | 4
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (4.4) |  | 52.5 (4.4)
Gender [Number; unit: participants]
  Female | 1 |  | 1
  Male | 3 |  | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Urine Sodium Excretion
Description: Within-subject comparison of increase in urine sodium excretion following saline loading before RSD and 13 weeks following RSD.
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected, endpoints not measured
Arm/Group | Early Renal Denervation | Late Renal Denervation
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Urine Volume
Description: Urine volume following furosemide therapy after sodium loading.
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Groups:
- Early Symplisity Renal Denervation: Subjects undergo Symplicity Renal Denervation within 2 weeks of baseline visit will follow usual care after week 13 visit
  Symplicity Renal Denervation: Renal denervation
- Late Symplisity Renal Denervation: Subjects following usual care until week 13 visit will then undergo Symplicity Renal Denervation within 2 weeks of Week 13 visit
  Symplicity Renal Denervation: Renal denervation
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: 24-hour Urine Sodium Excretion
Description: Difference in 24-hour urine sodium excretion, compared between pre-RSD and 13 weeks after RSD.
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Glomerular Filtration Rate
Description: Estimated Glomerular Filtration Rate (GFR) by creatinine and cystatin C
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Serum Cystatin C
Description: Study terminated early, endpoints not measured
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Blood Urea Nitrogen (BUN) Level
Description: Study terminated early, endpoints not measured
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Creatinine Clearance From 24-hour Urine Creatinine
Description: Study terminated early, endpoints not measured
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Urine Albumin
Description: Urine albumin
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Renal Resistive Index
Description: Intra-renal hemodynamics as measured by Renal Resistive Index (RRI) by renal Doppler ultrasonography Study terminated early, endpoints not measured
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Left Ventricular End Systolic Volume
Description: Echo: Left ventricular end systolic volume Study terminated early, endpoints not measured
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Left Ventricular Ejection Fraction
Description: Echo: Left Ventricular Ejection Fraction Study terminated early, endpoints not measured
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Global Longitudinal Strain
Description: Echo: Global longitudinal strain Study terminated early, endpoints not measured
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: LV End Systolic Dimension (LVESd)
Description: Echo: LV end systolic dimension (LVESd)
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: LV End Diastolic Dimension (LVEDd)
Description: Echo: LV end diastolic dimension (LVEDd)
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Left Atrial Size
Description: Echo: Left Atrial size
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Plasma N-terminal Pro-brain Natriuretic Peptide
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Resting Plasma Norepinephrine
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Resting Urine Norepinephrine
Time Frame: 13 Weeks following Renal Denervation
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Plasma Renin Activity
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Plasma Aldosterone
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: 6 Minute Walk Test
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire Score
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Patient Global Assessment
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Symplisity Renal Denervation | Late Symplisity Renal Denervation
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: New York Heart Association (NYHA) Functional Classification
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Renal Denervation | Late Renal Denervation
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Heart Rate Variability
Description: Heart rate variability indices by Holter
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Renal Denervation | Late Renal Denervation
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Tissue Doppler Indices
Description: Echo: Tissue Doppler indices
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Renal Denervation | Late Renal Denervation
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Left Ventricular End Diastolic Volume
Description: Echo: Left Ventricular End Diastolic Volume
Time Frame: 13 Weeks following Renal Denervation
Population: Study terminated early, data not collected and therefore endpoints were not measured.
Arm/Group | Early Renal Denervation | Late Renal Denervation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to one year post randomization
Arm/Group | Early Renal Denervation | Late Renal Denervation
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/0
Other Adverse Events (participants affected / at risk) | 1/4 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Renal Denervation (N=4) | Late Renal Denervation (N=0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Renal Denervation (N=4) | Late Renal Denervation (N=0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Non Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Data Safety Monitoring Board (DSMB) terminated trial based upon noted lack of efficacy in manufacturers pivotal trials. Endpoint data not collected or analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No